CLINICAL TRIAL: NCT02335645
Title: AlterG ACL Return to Running Case Series
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Physical Therapist, Nationwide Children's Hospital
Other Study IDs: IRB14-00823
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: ACL reconstruction; Running Mechanics; Physical Therapy; Knee; Video Analysis; Body Weight Supported Treadmill

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Body Weight Supported Treadmill: Post surgical ACL patients who will complete standard ACL protocol with the addition of body weight supported treadmill use.
  Interventions: Other: Body Weight Supported Treadmill Use of Patients with ACL Reconstruction

INTERVENTIONS:
Other: Body Weight Supported Treadmill Use of Patients with ACL Reconstruction — Standard ACL protocol will be followed throughout the treatment of each patient. The only variance from treatment will be using body weight supported treadmill and video gait analysis to help guide treatment.
  The first analysis will be performed at week 6 after surgery. Motion capture sensors will be placed on the patient at different anatomical positions. The patient will then run in a body weight supported treadmill. During this run, video capture will be performed and later analyzed to determine biomechanical kinematics.
  Based on findings of video gait analysis, exercise progression will be altered to improve deficits found. This process will be repeated at week 8 of rehabilitation in the body weight supported treadmill.
  At week 10 and 12, the patient will shift treatment from the body weight supported treadmill, to a standard treadmill. The process will be repeated using the same anatomical landmarks and video capture.

SUMMARY:
This case series will follow standard ACL protocol, while using biomechanical movement analysis to analyze running mechanics using a body weight supported treadmill.

Standard ACL protocol will be followed throughout the treatment of each patient. The only variance from treatment will be using motion analysis software to analyze gait patterns at different points throughout the rehabilitation.

The first motion analysis will be performed at week 6 of the rehabilitation process. Prior to this treatment, manual muscle testing of the hip, knee and ankle using a handheld dynamometer, two outcome measures, range of motion, pain, and patient satisfaction will be performed. At this treatment, motion capture sensors will be placed on the patient at different anatomical positions. The patient will then run in a body weight supported treadmill. During this run, video capture will be performed and later analyzed to determine biomechanical kinematics.

This process will be repeated at week 8 of rehabilitation in the body weight supported treadmill.

At week 10, the patient will shift treatment from the body weight supported treadmill, to a standard treadmill. The process will be repeated using the same anatomical landmarks and video capture.

The final video capture will be performed at week 12. At this visit, video capture will be performed. The patient will also repeat all test, measures, and questionnaires from week 6.

At all visits between video capturing, standard PT will be performed with a focus on patient deficits and following the standard protocol.

DETAILED DESCRIPTION:
Each year, up to 250,000 Anterior Cruciate Ligament (ACL) reconstructions are performed in the United States.(1) Individuals who undergo ACL reconstruction vary from the weekend warrior to high level professional athletes. With a majority of ACL injuries occurring from a sports injury, returning to running is a key portion of the rehabilitation process.(2) Following an ACL tear, knee laxity and instability are a common complaint. Due to this, individuals are classified as coper or non-copers.(3) Copers are individuals who are able to maintain their previous function with conservative treatment. Non-copers are persons who are unable to return to their previous level of activity due to instability or who perform high level activities. Non-copers will undergo ACL reconstruction surgery, followed by a lengthy rehabilitation process.(3)

With extensive knowledge on running mechanics, it is important to consider these normal mechanics following ACL surgery.(4, 5) Following ACL surgery and rehabilitation, several variances in gait pattern are known to exist for 6 months or greater. Several Studies have demonstrated abnormal knee torques following ACL surgery for well over 6 months.(6) With known deficits lasting for several months, we must consider these mechanics and return to sport criteria when returning an athlete to sports competition. With the highest risk of reinjury in the first several months, understanding gait mechanics and risk factors is vital to a successful ACL rehabilitation.(6) As a clinician, the most important aspect to consider a rehabilitation successful is an athlete's full return to the sport or activity of their choice, at the highest level. In order to do this, we must understand all areas of their mechanics and limit any deficits throughout the process.

Over time, ACL protocols have progressively changed from a standard conservative plan, to an accelerated protocol, with return to running at around 6 months.(7) This is nearly twice as fast as the conservative plan. As the time to return to sports participation continues to decrease, understanding mechanics and correcting deficits is important to an overall successful surgery, rehabilitation, and patient. The ability to progressively decrease treatment times has been made possible by increased knowledge and ever improving technology.

One piece of technology that allows this decrease in rehabilitation time is the use of a body weight supported treadmill to allow a much quicker return to running, within the limitations of a protocol. One such example is the AlterG, Anti-Gravity treadmill. This treadmill allows a patient to run with as little as 20% of their body weight using an air pressure system for unweighting. This type of unweighting allows for safe and normal gait mechanics, in a pain free system. This type of treadmill also allows a clinician to adjust and monitor changes and improvements as a patient progresses through a treatment.(8)

The purpose of this case series is to assess the novel treatment of body weight supported treadmill use early in the rehabilitation protocol to address running deficits and mechanics within the standard of care.

The primary objectives are to determine if early running with the use of body weight support, result in decreased pain and higher feelings of success early in the rehabilitation process. The secondary objective of this study is to determine if running mechanics are altered with the use of body weight support, following ACL reconstruction surgery.

This is a single site study to be performed at the Westerville Close to Home Sports Physical Therapy Location.

This is a case series to assess the running mechanics following ACL surgery using both standard and body weight supported treadmill. Patients who are referred to Westerville following an ACL reconstruction surgery will be offered the opportunity to participate in this study. Patients will begin their standard protocol for the first 3-4 weeks before being approached to participate in this study. At this time, if they are progressing well through their protocol, they will be approached and asked if they would like information regarding this study. After explaining the study and answering any patient or parent questions, informed consent and assent will be obtained for those individuals wishing to participate. The participants will be screened to see if they meet the inclusion criteria at this time. If the patient meets the criteria and is agreeable to participate in this study, standard protocol will continue to be followed until week six. Standard care will continue for all treatments excepts four visits, occuring during weeks 6,8,10,and 12, where a video recording of running gait mechanics will be performed to analysis biomechanics throughout the rehabilitation process.

At week 6, pretreatment evaluation measures will be performed. These will consist of:

* Pediatric International Knee Document Committee (Pedi-IKDC) is a self-reported questionnaire relating to a young patients function, symptoms, and sports activity. This is a valid study in patients ages 10-18. (1)
* Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient reported outcome measure intended for use in knee injuries that may result in osteoarthritis such as anterior cruciate reconstruction. This measure is valid in individual's age 13-79 years and consists of 5 subscales. (2)
* The use of the Numerical Pain Rating Scale (NPRS) for assessing pain has been validated for use in adolescent patients and has been found to have a minimal detectable change of 2 points. The NPRS will be administered at the beginning and end of every treatment session. (3)
* Manual Muscle Testing (MMT) will be administered using a hand held dynamometer. This will be performed for hip flexion, extension, abduction and adduction. MMT will also be performed for knee flexion and extension, as well ankle plantar flexion, dorsiflexion, inversion, and eversion. (4)
* Range of Motion Testing well also be completed at this time, measuring all hip, knee and ankle movements.

Treatment interventions will start with the recording of gait mechanics during the use of the AlterG body weight supported treadmill.

Following the pretreatment evaluation, the patient will prepare to use the body weight supported treadmill. The patient will wear the appropriate shorts associated with the treadmill based on waist size. At this time, reflective markers will be placed on anatomical position. The marker positions will include: Tibial tuberosity, mid patella, anterior mid thigh, lateral mid thigh, lateral knee joint line, lateral malleoli, fibula head, lateral calcaneus, lateral fifth metatarsal head, lumbar spine (L3) and iliac crest. These markers will later be used with the mechanics analysis software to determine running biomechanics. After the markers are in place, the patient will enter the AlterG body weight supported treadmill. After the treadmill calibrates, they will begin the first walk-jog progression. The following setting will be used for the first run based on standard protocol.

* 60% Body weight
* 1 minute walk/2 minute jog (repeated 3 times)
* 1% incline
* Walk: 3.0mph
* Run: Desired speed of choice

After completion, markers will be removed and the patient will begin standard physical therapy (PT) care per protocol.

Standard PT care will be continued from weeks 6-8 with a focus on patient deficits and progression per protocol. Patient will continue to use the AlterG treadmill but will not be recorded at this time. The AlterG setting will be continually progressed as able.

At 8 weeks, the patient will again be record in the AlterG body weight supported treadmill. The patient will get prepared to use the body weight supported treadmill. The patient will wear the appropriate shorts associated with the treadmill based on waist size. At this time, reflective markers will be placed on anatomical position. These markers will later be used with the mechanics analysis software to determine running biomechanics. After the markers are in place, the patient will enter the AlterG body weight supported treadmill. After the treadmill calibrates, they will begin the first walk-jog progression. The following setting will be used for the first run based on standard protocol.

* 75% Body weight
* 1 minute walk/4 minute jog (repeated 3 times)
* 1% incline
* Walk: 3.0mph
* Run: Desired speed of choice

Standard physical therapy care will be continued from weeks 8-10 with a focus on patient deficits and progression per protocol. Patient will continue to use the AlterG treadmill but will not be recorded at this time.

At 10 weeks, the patient will again be recorded but treadmill use will be changed to a standard treadmill with no body weight support. At this time, reflective markers will be placed on anatomical position. These markers will later be used with the mechanics analysis software to determine running biomechanics. After the markers are in place, the patient will begin running on the treadmill per standard protocol. The following setting will be used for the first run on the standard treadmill based on standard protocol.

* 1 minute walk/2 minute jog (repeated 3 times)
* 1% incline
* Walk: 3.0mph
* Run: Desired speed of choice

Standard PT care will be continued from weeks 10-12 with a focus on patient deficits and progression per protocol. Patient will continue to use the standard treadmill but will not be recorded at this time.

At 12 weeks, the patient will again be recorded in a standard treadmill with no body weight support. At this time, reflective markers will be placed on anatomical position. These markers will later be used with the mechanics analysis software to determine running biomechanics. After the markers are in place, the patient will begin running on the treadmill per standard protocol. The following setting will be used for the first run on the standard treadmill based on standard protocol.

* 1 minute walk/ 5 minute jog (repeated 3 times)
* 1% incline
* Walk: 3.0mph
* Run: Desired speed of choice

Following the 4th recording, the patient will be completed with the research study. The patient will again repeat all outcome measures and pretreatment testing at this time. Testing will include:

* Knee Osteoarthritis Outcome Score
* Pediatric International Knee Disability Committee
* Manual muscle testing with the use of hand held dynamometer
* Range of motion with the use of a goniometer
* Functional testing will also be performed at this time. Following 12 weeks of therapy, functional testing is typically done to assess progress. Functional testing at this time will include three different tests:
* Single Leg hop test:
* Triple Hop Test:
* Triple Crossover Hop Test:

At that time, standard care will continue with possible discharge to functional rehabilitation or continuing PT care based on their progress and functional status.

Throughout all standard visits, patients will be seen for 45-90 minutes 2 times per week. Treatment times will vary as the patient progresses through the rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of post operative anterior cruciate reconstruction surgery.

Exclusion Criteria:

* Patient has concurrent diagnosis of meniscal repair with ACL surgery.
* Patient ACL surgery is apophyseal sparing.
* Patient is unable to follow directions
* History of activity limiting illness
* Inability to attend follow up appointments
* Current Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will include post operative ACL patients who meet the eligibility criteria who are being treated at Nationwide Children's Westerville Physical Therapy location.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Pedi-IKDC | Measure week 6 and week 12 following surgery
  Pediatric International Knee Document Committee (Pedi-IKDC) is a self-reported questionnaire relating to a young patients function, symptoms, and sports activity. This is a valid study in patients ages 10-18
Change in KOOS | Measure week 6 and week 12 following surgery
  Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient reported outcome measure intended for use in knee injuries that may result in osteoarthritis such as anterior cruciate reconstruction. This measure is valid in individual's age 13-79 years and consists of 5 subscales
Change in numeric pain rating scale | Measure week 6 and week 12 following surgery
  The use of the Numerical Pain Rating Scale (NPRS) for assessing pain has been validated for use in adolescent patients and has been found to have a minimal detectable change of 2 points. The NPRS will be administered at the beginning and end of every treatment session
Change in manual muscle testing | Measure week 6 and week 12 following surgery
  Manual Muscle Testing (MMT) will be administered using a hand held dynamometer. This will be performed for hip flexion, extension, abduction and adduction. MMT will also be performed for knee flexion and extension, as well ankle plantar flexion, dorsiflexion, inversion, and eversion.

SECONDARY OUTCOMES:
Change in dynamic knee valgus | Measured week 6 and week 12 following surgery
  Reflective markers will be placed at anterior mid thigh, middle patella, and tibial tuberosity. These markers will be analyzed using video analysis to measure knee valgus throughout gait.
Change in dynamic knee flexion | Measured week 6,8,10,12 following surgery
  Reflective markers will be placed at lateral mid thigh, lateral knee joint line, and lateral malleolus . These markers will be analyzed using video analysis to measure knee valgus throughout gait.
Change in ankle dorsiflexion/plantar flexion | Measured week 6,8,10, and 12 following surgery
  Reflective markers will be placed at fibular head, lateral calcaneus, and lateral fifth metatarsal head . These markers will be analyzed using video analysis to measure knee valgus throughout gait.
Change in vertical excursion | measured week 6,8,10,12 following surgery
  Reflective marker will be placed on the lumbar spine L3 process. These markers will be analyzed using video analysis to measure knee valgus throughout gait.
change in hip drop | measured week 6,8,10,12 following surgery
  Reflective markers will be placed on bilateral iliac crest. These markers will be analyzed using video analysis to measure knee valgus throughout gait.
Change in stride length | measured week 6,8,10,12 following surgery
  Video analysis will be used to measure stride length bilaterally during gait.
Change in cadence | measured week 6,8,10,12 following surgery
  Video analysis will be used to measure cadence during gait.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital Sports and Ortho PT Westerville, Westerville, Ohio, United States